CLINICAL TRIAL: NCT00072761
Title: Silent Cerebral Infarct Transfusion Multi-Center Clinical Trial
Acronym: SIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Michael DeBaun, Professor or Pediatrics and Medicine, JC Peterson Endowed Chair, Vice Chair of Clinical Research, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NS42804; 5U01NS042804-07 (NIH)
Record Dates: First submitted 2003-11-10; First posted 2003-11-13 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Sickle Cell Anemia; Stroke
Keywords: silent cerebral infarct; silent stroke; sickle cell anemia; stroke; transfusion therapy
MeSH Terms: conditions — Anemia, Sickle Cell; Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transfusion Group (Active Comparator): Participants allocated to the transfusion arm will receive blood transfusion therapy every 4-6 weeks for 36 months.
  Interventions: Procedure: transfusion therapy
- Observation Group (No Intervention): Participants allocated to the observation arm will be treated according to standard care and will receive a quarterly physical examination by a study hematologist for 36 months.

INTERVENTIONS:
Procedure: transfusion therapy — Those in the blood transfusion group will receive at least monthly blood transfusion therapy.
  Arms: Transfusion Group

SUMMARY:
The goal of this study is to determine the effectiveness of blood transfusion therapy for prevention of silent cerebral infarct (stroke) in children with sickle cell anemia.

DETAILED DESCRIPTION:
Silent cerebral infarct (stroke) is the most common cause of severe cognitive impairments and related neurological functions in children with sickle cell anemia. Currently there exists no systemic strategy to identify or treat children with silent strokes.

The primary aim of this trial is to determine the effectiveness of blood transfusion therapy for the prevention of silent strokes in children with sickle cell anemia. This trial will also determine if blood transfusion therapy will prevent further cerebral injury and if the measured benefits of the therapy outweigh the risks associated with it.

Participants in this multi-center trial will be randomly assigned to one of 2 groups-the blood transfusion group or the observation group. Those in the blood transfusion group will receive at least monthly blood transfusion therapy. All participants will have history and physical examinations every 3 months, and magnetic resonance imaging (MRI) at the beginning of their entry into the study and at study exit.

Advances in the understanding and treatment of silent strokes will likely lead to a decrease in the burden associated with cerebral injury in children with sickle cell anemia and change the standard care for these children.

Statistical Analyses: The original statistical analysis plan suggested a simple difference in proportions between the proportion of individuals with an endpoint in the transfusion group and the proportion of individuals with an endpoint in the usual care group using a traditional chi squared test. The data should be analyzed according to an intent to treat principal. Because of various logistical concerns in SIT, some individuals were not imaged within the 36-month window (30-42 months). We propose using all available information by changing the primary analysis from a dichotomous (yes/no) endpoint to a traditional epidemiological endpoint of an incidence rate in the group randomized to transfusion to the incidence rate in the group randomized to usual care. We will compute the incidence ratio:

(a/ta)/(b/tb)

Where "a" is the number of endpoints in the transfusion group, "ta" is the sum of the individual times at risk of the individuals randomized to the transfusion group, "b" is the number of endpoints in the observation group and "tb" is the sum of the individual times at risk of the individuals randomized to the observation group.

Since the standard statistical test for it being different than 1.0 involves the assumption of a Poisson distribution, we will compute an "exact" 95% confidence interval using a bootstrap with a large number of replications.

ELIGIBILITY:
INCLUSION:

* Patient must have sickle cell anemia (hemoglobin SS) or sickle beta thalassemia (hemoglobin SB) as confirmed at the local institution.
* Participating institutions must submit documentation of the diagnostic hemoglobin analysis to the Statistical and Clinical Coordinating Centers to confirm the diagnosis of sickle cell anemia prior to randomization.
* Patient must be 5 through 14 years of age.
* Patient must have a cerebral infarct documented by MRI scan as read by the neuroradiology panel.
* Informed consent with assent in accordance with the institutional policies (institutional Institutional Review Board approval) and Federal guidelines (approved by the United States Department of Health and Human Services) must be signed by the patient's legally authorized guardian acknowledging written consent to join the study. When suitable, patients will be requested to give their assent to join the study.

EXCLUSION:

* Patient with a history of a focal neurologic event lasting more than 24 hours with medical documentation or a history of prior overt stroke.
* Patients with a transcranial doppler (TCD) study with a time-averaged mean velocity greater than 200 cm/sec verified by the study radiologist.
* Patients with other neurological problems, such as neurofibromatosis, lead poisoning, or tuberous sclerosis.
* Patients with HIV infection.
* Pregnancy.
* Patients who received treatment with anti-sickling drugs or hydroxyurea within 3 months or anticipate receiving anti-sickling drugs or hydroxyurea during the course of the study.
* Abnormal kidney function (creatinine > 2x upper limit of normal).
* Patients on chronic blood transfusion therapy for other reasons.
* Patients judged not likely to be compliant by his/her hematologist and local nurse coordinator based on previous compliance in clinic appointments and following advice. Specifically, families that have missed at least two appointments without notification within 12 months prior to the trial or parents of potential patients that have been reported for medical or education neglect are not eligible for this trial.
* Patients unable to receive blood transfusion because of alloimmunization.
* Patients with permanent or semi-permanent metallic (braces on teeth) structures attached to their body. Such patients cannot obtain a MRI of the head to assess the presence of silent cerebral infarcts.
* Siblings randomized in the trial.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Actual)
Dates: Start 2004-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. DeBaun, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Buchanan GR, DeBaun MR, Quinn CT, Steinberg MH. Sickle cell disease. Hematology Am Soc Hematol Educ Program. 2004:35-47. doi: 10.1182/asheducation-2004.1.35. PMID 15561675
- [Background] Vendt BA, McKinstry RC, Ball WS, Kraut MA, Prior FW, Barton B, Casella JF, DeBaun MR. Silent Cerebral Infarct Transfusion (SIT) trial imaging core: application of novel imaging information technology for rapid and central review of MRI of the brain. J Digit Imaging. 2009 Jun;22(3):326-43. doi: 10.1007/s10278-008-9114-3. Epub 2008 Apr 9. PMID 18398653
- [Background] Casella JF, King AA, Barton B, White DA, Noetzel MJ, Ichord RN, Terrill C, Hirtz D, McKinstry RC, Strouse JJ, Howard TH, Coates TD, Minniti CP, Campbell AD, Vendt BA, Lehmann H, Debaun MR. Design of the silent cerebral infarct transfusion (SIT) trial. Pediatr Hematol Oncol. 2010 Mar;27(2):69-89. doi: 10.3109/08880010903360367. PMID 20201689
- [Background] Jordan LC, McKinstry RC 3rd, Kraut MA, Ball WS, Vendt BA, Casella JF, DeBaun MR, Strouse JJ; Silent Infarct Transfusion Trial Investigators. Incidental findings on brain magnetic resonance imaging of children with sickle cell disease. Pediatrics. 2010 Jul;126(1):53-61. doi: 10.1542/peds.2009-2800. Epub 2010 Jun 14. PMID 20547639
- [Background] Bhatnagar P, Purvis S, Barron-Casella E, DeBaun MR, Casella JF, Arking DE, Keefer JR. Genome-wide association study identifies genetic variants influencing F-cell levels in sickle-cell patients. J Hum Genet. 2011 Apr;56(4):316-23. doi: 10.1038/jhg.2011.12. Epub 2011 Feb 17. PMID 21326311
- [Background] Jordan LC, Casella JF, DeBaun MR. Prospects for primary stroke prevention in children with sickle cell anaemia. Br J Haematol. 2012 Apr;157(1):14-25. doi: 10.1111/j.1365-2141.2011.09005.x. Epub 2012 Jan 9. PMID 22224940
- [Background] DeBaun MR, Sarnaik SA, Rodeghier MJ, Minniti CP, Howard TH, Iyer RV, Inusa B, Telfer PT, Kirby-Allen M, Quinn CT, Bernaudin F, Airewele G, Woods GM, Panepinto JA, Fuh B, Kwiatkowski JK, King AA, Rhodes MM, Thompson AA, Heiny ME, Redding-Lallinger RC, Kirkham FJ, Sabio H, Gonzalez CE, Saccente SL, Kalinyak KA, Strouse JJ, Fixler JM, Gordon MO, Miller JP, Noetzel MJ, Ichord RN, Casella JF. Associated risk factors for silent cerebral infarcts in sickle cell anemia: low baseline hemoglobin, sex, and relative high systolic blood pressure. Blood. 2012 Apr 19;119(16):3684-90. doi: 10.1182/blood-2011-05-349621. Epub 2011 Nov 17. PMID 22096242
- [Background] Thangarajh M, Yang G, Fuchs D, Ponisio MR, McKinstry RC, Jaju A, Noetzel MJ, Casella JF, Barron-Casella E, Hooper WC, Boulet SL, Bean CJ, Pyle ME, Payne AB, Driggers J, Trau HA, Vendt BA, Rodeghier M, DeBaun MR. Magnetic resonance angiography-defined intracranial vasculopathy is associated with silent cerebral infarcts and glucose-6-phosphate dehydrogenase mutation in children with sickle cell anaemia. Br J Haematol. 2012 Nov;159(3):352-9. doi: 10.1111/bjh.12034. Epub 2012 Sep 7. PMID 22958163
- [Background] Quinn CT, McKinstry RC, Dowling MM, Ball WS, Kraut MA, Casella JF, Dlamini N, Ichord RN, Jordan LC, Kirkham FJ, Noetzel MJ, Roach ES, Strouse JJ, Kwiatkowski JL, Hirtz D, DeBaun MR. Acute silent cerebral ischemic events in children with sickle cell anemia. JAMA Neurol. 2013 Jan;70(1):58-65. doi: 10.1001/jamaneurol.2013.576. PMID 23108767
- [Background] Bean CJ, Boulet SL, Ellingsen D, Pyle ME, Barron-Casella EA, Casella JF, Payne AB, Driggers J, Trau HA, Yang G, Jones K, Ofori-Acquah SF, Hooper WC, DeBaun MR. Heme oxygenase-1 gene promoter polymorphism is associated with reduced incidence of acute chest syndrome among children with sickle cell disease. Blood. 2012 Nov 1;120(18):3822-8. doi: 10.1182/blood-2011-06-361642. Epub 2012 Sep 10. PMID 22966170
- [Background] Milton JN, Sebastiani P, Solovieff N, Hartley SW, Bhatnagar P, Arking DE, Dworkis DA, Casella JF, Barron-Casella E, Bean CJ, Hooper WC, DeBaun MR, Garrett ME, Soldano K, Telen MJ, Ashley-Koch A, Gladwin MT, Baldwin CT, Steinberg MH, Klings ES. A genome-wide association study of total bilirubin and cholelithiasis risk in sickle cell anemia. PLoS One. 2012;7(4):e34741. doi: 10.1371/journal.pone.0034741. Epub 2012 Apr 27. PMID 22558097
- [Background] DeBaun MR, Armstrong FD, McKinstry RC, Ware RE, Vichinsky E, Kirkham FJ. Silent cerebral infarcts: a review on a prevalent and progressive cause of neurologic injury in sickle cell anemia. Blood. 2012 May 17;119(20):4587-96. doi: 10.1182/blood-2011-02-272682. Epub 2012 Feb 21. PMID 22354000
- [Background] Glassberg JA, Wang J, Cohen R, Richardson LD, DeBaun MR. Risk factors for increased ED utilization in a multinational cohort of children with sickle cell disease. Acad Emerg Med. 2012 Jun;19(6):664-72. doi: 10.1111/j.1553-2712.2012.01364.x. PMID 22687181
- [Background] An P, Barron-Casella EA, Strunk RC, Hamilton RG, Casella JF, DeBaun MR. Elevation of IgE in children with sickle cell disease is associated with doctor diagnosis of asthma and increased morbidity. J Allergy Clin Immunol. 2011 Jun;127(6):1440-6. doi: 10.1016/j.jaci.2010.12.1114. Epub 2011 Mar 9. PMID 21388662
- [Result] DeBaun MR, Gordon M, McKinstry RC, Noetzel MJ, White DA, Sarnaik SA, Meier ER, Howard TH, Majumdar S, Inusa BP, Telfer PT, Kirby-Allen M, McCavit TL, Kamdem A, Airewele G, Woods GM, Berman B, Panepinto JA, Fuh BR, Kwiatkowski JL, King AA, Fixler JM, Rhodes MM, Thompson AA, Heiny ME, Redding-Lallinger RC, Kirkham FJ, Dixon N, Gonzalez CE, Kalinyak KA, Quinn CT, Strouse JJ, Miller JP, Lehmann H, Kraut MA, Ball WS Jr, Hirtz D, Casella JF. Controlled trial of transfusions for silent cerebral infarcts in sickle cell anemia. N Engl J Med. 2014 Aug 21;371(8):699-710. doi: 10.1056/NEJMoa1401731. PMID 25140956
- [Derived] Hsu P, Gay JC, Lin CJ, Rodeghier M, DeBaun MR, Cronin RM. Economic evaluation of regular transfusions for cerebral infarct recurrence in the Silent Cerebral Infarct Transfusion Trial. Blood Adv. 2021 Dec 14;5(23):5032-5040. doi: 10.1182/bloodadvances.2021004864. PMID 34607344
- [Derived] Dowling MM, Noetzel MJ, Rodeghier MJ, Quinn CT, Hirtz DG, Ichord RN, Kwiatkowski JL, Roach ES, Kirkham FJ, Casella JF, DeBaun MR. Headache and migraine in children with sickle cell disease are associated with lower hemoglobin and higher pain event rates but not silent cerebral infarction. J Pediatr. 2014 May;164(5):1175-1180.e1. doi: 10.1016/j.jpeds.2014.01.001. Epub 2014 Feb 13. PMID 24529619
- [Derived] Savage WJ, Barron-Casella E, Fu Z, Dulloor P, Williams L, Crain BJ, White DA, Jennings JM, Van Eyk JE, Debaun MR, Everett A, Casella JF. Plasma glial fibrillary acidic protein levels in children with sickle cell disease. Am J Hematol. 2011 May;86(5):427-9. doi: 10.1002/ajh.21995. PMID 21523806
- [Derived] Williams LM, Fu Z, Dulloor P, Yen T, Barron-Casella E, Savage W, Van Eyk JE, Casella JF, Everett A. Hemoglobin depletion from plasma: considerations for proteomic discovery in sickle cell disease and other hemolytic processes. Proteomics Clin Appl. 2010 Dec;4(12):926-30. doi: 10.1002/prca.201000054. PMID 21179892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in December, 2004 and ended May, 2010. Among the 1074 children screened with a MRI of the brain, 1.9% (20 of 1074) had strokes and 35.2% (379 of 1074) had infarct-like lesions. 196 participants completed all pre-randomization procedures and were successfully randomly allocated.
Groups:
- Transfusion Group: The transfusion group received blood transfusion therapy every 4-6 weeks for 36 months.
- Observation Group: The observation group received standard care therapy and quarterly physical examination by a study hematologist for 36 months.
Period: Overall Study
Arm/Group | Transfusion Group | Observation Group
Started | 99 | 97
Completed | 90 | 95
Not Completed | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transfusion Group | Observation Group | Total
Number analyzed (Participants) | 99 | 97 | 196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 99 | 97 | 196
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 10 [5 to 15] | 10 [5 to 15] | 10 [5 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 45 | 85
  Male | 59 | 52 | 111
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 91 | 90 | 181
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of an Infarct, Defined as a Stroke or a New or Enlarged Silent Cerebral Infarct
Description: The primary end point was the recurrence of infarct or hemorrhage as determined by neuroimaging, clinical evidence of permanent neurologic injury, or both. A new infarct had to meet the criteria for a silent cerebral infarction; an enlarged silent cerebral infarct was defined as a previously identified silent cerebral infarct that increased by at least 3 mm along any linear dimension in any plane on MRI.
Time Frame: From study entry to study exit
Population: Randomization assignments were provided by the statistical data coordinating center with the use of a permuted block design, with stratification according to site, age, and sex. Participants were assigned in a 1:1 ratio to the observation or transfusion group and were followed until study exit or study endpoint.
Measure: Number; unit: infarct recurrence per 100 person years
Arm/Group | Transfusion Group | Observation Group
Number analyzed (Participants) | 99 | 97
infarct recurrence per 100 person years | 2.0 | 4.8

ADVERSE EVENTS:
Arm/Group | Transfusion Group | Observation Group
Serious Adverse Events (participants affected / at risk) | 6/99 | 16/97
Other Adverse Events (participants affected / at risk) | 99/99 | 97/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transfusion Group (N=99) | Observation Group (N=97)
Stroke (General disorders) | 1 | 7
Silent Cerebral Infarct (General disorders) | 5 | 7
Transient Ischemic Attack (General disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Transfusion Group (N=99) | Observation Group (N=97)
Vaso-Occlusive Pain (General disorders) | 32 (126) | 56 (295)
Acute Chest Syndrome (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 24 (41)
Priapism (General disorders) | 1/59 (1) | 7/52 (10) — This event was documented in male participants only.
Symptomatic avascular necrosis of the hip (General disorders) | 1 (1) | 6 (6)
Headache (General disorders) | 24 (76) | 30 (93)
Blood-transfusion reaction (General disorders) | 15/90 (24) | 1/31 (1)
Ferritin > 1500 ng/ml (General disorders) | 76/90 (1479) | 3/31 (33)

LIMITATIONS AND CAVEATS:
The SIT Trial results are not directly applicable to all children with SCA. Those who were on hydroxyurea therapy for severe disease, had abnormally elevated TCDs, were receiving blood transfusion for stroke prevention or had epilepsy were excluded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No